CLINICAL TRIAL: NCT06596122
Title: The Effect of Vitamin D Supplementation in Breast Cancer Patients Receiving Taxane-based Chemotherapy
Brief Title: Vitamin D Supplementation in Breast Cancer Patients
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Abdelrahman Mahmoud (Other)
Responsible Party: Sponsor-Investigator, Abdelrahman Mahmoud, Dr, Cairo University
Organization: Cairo University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Vitamin D in cancer patients
Record Dates: First submitted 2024-09-11; First posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Peripheral Neuropathic Pain
Keywords: Cholecalciferol; Breast cancer; Neuropathic pain; Taxane; Paclitaxel; Vitamin D3
MeSH Terms: conditions — Breast Neoplasms; Neuralgia | interventions — Cholecalciferol

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: Only the neurologist conducting the Modified Total Neuropathy Score (mTNS) assessment will be blinded.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Intervention group (Active Comparator): In conjunction with the AC-T chemotherapy protocol, individuals in the intervention group who have a vitamin D deficiency will receive vitamin D replacement therapy.
  Interventions: Drug: Vitamin D (Cholecalciferol )
- The control group (No Intervention): only the standard of care will be administered.

INTERVENTIONS:
Drug: Vitamin D (Cholecalciferol ) — In conjunction with the AC-T chemotherapy protocol, individuals in the intervention group who have a vitamin D deficiency will receive an oral loading dose of 50,000 IU weekly for eight weeks. Subsequently, they will be given 100,000 IU monthly until the completion of their chemotherapy treatment.
  Arms: Intervention group

SUMMARY:
It is a randomized clinical trial aimed at exploring the neuroprotective effect of vitamin D3 (Cholecalciferol) supplementation in conjunction with paclitaxel-based chemotherapy among breast cancer patients with vitamin D insufficiency or deficiency.

DETAILED DESCRIPTION:
This study is a two-arm randomized controlled trial with 132 participants, evenly randomized into an intervention group and a control group. Both groups are scheduled to receive Adriamycin-Cyclophosphamide followed by paclitaxel (AC-T) chemotherapy protocol. The intervention group will undergo paclitaxel-based chemotherapy, along with vitamin D replacement therapy. Conversely, the control group will follow the AC-T protocol without the addition of vitamin D replacement therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Female aged 18 to 65 years old.
2. Histologically confirmed breast cancer.
3. Eastern Cooperative Oncology Group (ECOG) performance status of less than or equal to 2 [21] [22].
4. All patients should fulfill the criteria of the initiation of taxane-based chemotherapy such as absolute neutrophil count (ANC) > 1,500/mcL, platelets > 100,000/mcL, hemoglobin ≥ 9 g/mL, Aspartate Aminotransferase (AST) (Serum Glutamic-Oxaloacetic Transaminase) (SGOT) to Alanine Aminotransferase (ALT), (Serum Glutamic-Pyruvic Transaminase) (SGPY) ratio (AST (SGOT)/ALT (SGPT)) < 2.5 x institutional upper limit of normal (ULN), total bilirubin less than or equal to 1.5 x institutional ULN, serum creatinine < 1.5 x institutional ULN.
5. Stage I-III breast cancer scheduled to undergo adjuvant or neoadjuvant paclitaxel-based chemotherapy for breast cancer using doxorubicin 60 mg/m² and cyclophosphamide 600 mg/m² followed by paclitaxel 80 mg/m² weekly for 12 weeks protocol code BRAJACTW [23].
6. Vitamin D insufficiency defined as serum level < 30 ng/ml.
7. Ability to give informed consent as per the legal requirement.

Exclusion Criteria:

1. Prior neurotoxic chemotherapy including paclitaxel.
2. Metastatic carcinoma.
3. History of any other malignancy except malignancy that was treated with curative intent and for which there has been no known active disease for more than 3 years prior to randomization, curatively treated non-melanoma skin malignancy, cervical cancer in situ, in situ ductal carcinoma, or breast in situ lobular carcinoma.
4. Grade II neuropathy or higher based on the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0. neurosensory or neuromotor neuropathy, regardless of causality.
5. Patients who are scheduled to receive any neurotoxic chemotherapeutic agents such as platinum compounds (carboplatin, cisplatin), vinorelbine, eribulin, and ixabepilone.
6. Diabetes mellitus
7. Psychiatric disorders that limit ability to comply with study protocol i.e., history of regular exacerbation of major psychosis (schizophrenia, bipolar disorder) in last 2 years.
8. Known Fibromyalgia
9. Gastric bypass surgery.
10. Patients with chronic granuloma forming disorders (sarcoidosis or tuberculosis TB).
11. Known hyperparathyroidism.
12. Known thyroid dysfunction.
13. Known positive test for human immunodeficiency virus (HIV), hepatitis C virus, or acute or chronic hepatitis B infection.
14. Pregnancy and lactation.
15. Hypercalcemia (corrected blood calcium > 10.5 mg/dl or > 2.6 mmol/L)[24]
16. Hyperphosphatemia, serum phosphate concentration > 4.5 mg/dL [25]
17. History of symptomatic genitourinary stones within the past year.
18. Allergy to any cholecalciferol dosage form component.
19. Alcohol consumption.
20. Regular use of vitamin D > 2000 IU daily over the past year.
21. Inability to swallow pills.
22. Medications that may interfere with vitamin D metabolism, including enzyme inducing anticonvulsants, lithium, phenytoin, verapamil, orlistat, tuberculosis medications as isoniazid, and/or rifampin and estrogen-containing medications.
23. Patients receiving any of the following medications used to prevent CIPN: vitamin E, glutamine, nortriptyline, amitriptyline, tricyclic antidepressants, pregabalin, and duloxetine and other nutritional supplements as vitamin B during taxane administration.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 132 (Estimated)
Dates: Start 2024-10-15 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
The cumulative incidence and grading of paclitaxel-induced peripheral neuropathy (PIPN) | PIPN will be assessed throughout the 12-weeks paclitaxel administration phase.
  The incidence and grading of paclitaxel-induced peripheral neuropathy (PIPN) will be assessed using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) v5.0.

SECONDARY OUTCOMES:
The modified total neuropathy score mTNS. | The change in mTNS will be compared at weeks 18 and 24 relative to baseline.
  The Modified Total Neuropathy Score (mTNS) is a tool including six items that evaluate peripheral neuropathy symptoms by their presence, location, and characteristics, including sensory and motor symptoms, response to pinprick, vibration sensitivity, muscle strength, and deep tendon reflexes. Each item is scored on a scale from 0 to 4, with the total possible score ranging from 0 to 24. The sum of these scores yields a total score, with higher scores indicating more severe neuropathy.
EORTC QLQ-CIPN20 | Taxane-induced peripheral neuropathy using (EORTC QLQ-CIPN20) at weeks 13, 15,18, 21 and 24.
  The assessment of taxane-induced peripheral neuropathy will be carried out through interviews utilizing the Arabic version of the EORTC QLQ-CIPN20. This 20-item questionnaire, which includes sensory, motor, and autonomic subscales, will be employed for evaluations.
Quality of life | Quality of life (QOL) assessed at the first week, then at weeks 13 and 24.
  Quality of life (QOL) assessments will be conducted through interviews utilizing the Arabic version of the Functional Assessment of Cancer Therapy Breast Symptom Index (FBSI).

CONTACTS AND LOCATIONS:
Locations (1):
- Ain Shams University (El-Demerdash) Hospital, Cairo, Egypt